CLINICAL TRIAL: NCT03212144
Title: The Anti-Inflammatory Effects of Exercise and Peanut Consumption
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor enrollment
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Richard Sloan, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: #7466
Record Dates: First submitted 2017-06-08; First posted 2017-07-11 (Actual); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Peanut Consumption; High Intensity Aerobic Exercise
Keywords: nuts; exercise; vagal activity; peanuts; heart rate variability
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Data collection staff is masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training then Peanut Consumption (Experimental): Exercise group: 4 training sessions/week, 24 hour rest-periods between each training day. 3-min low intensity warm-up, and then exercise as rapidly as possible for 20 seconds, aiming to reach 85% of their maximum heart rate established during the submaximal cardiopulmonary exercise testing. Then followed by 40 seconds of low intensity exercise. Peanut group: Regular daily caloric intake estimated using data from 24hr recalls, the Miflin-St. Jeor equation, and stress/activity factors. Participants consume dry roasted, unsalted peanuts equivalent to approximately 10% of daily energy intake twice a day, range from approximately 2.4-3.6 ounces. Daily caloric intake will not differ from participants' typical diet. Participants are asked to bring back the empty, numbered peanut packets by the end of every week and will be given new packets weekly. Additionally, subjects will be informed that they will be randomly assessed weekly for compliance.
  Interventions: Other: High Intensity Interval Training
- Peanut Consumption then High Intensity Interval Training (Experimental): Exercise group: 4 training sessions/week, 24 hour rest-periods between each training day. 3-min low intensity warm-up, and then exercise as rapidly as possible for 20 seconds, aiming to reach 85% of their maximum heart rate established during the submaximal cardiopulmonary exercise testing. Then followed by 40 seconds of low intensity exercise. Peanut group: Regular daily caloric intake estimated using data from 24hr recalls, the Miflin-St. Jeor equation, and stress/activity factors. Participants consume dry roasted, unsalted peanuts equivalent to approximately 10% of daily energy intake twice a day, range from approximately 2.4-3.6 ounces. Daily caloric intake will not differ from participants' typical diet. Participants are asked to bring back the empty, numbered peanut packets by the end of every week and will be given new packets weekly. Additionally, subjects will be informed that they will be randomly assessed weekly for compliance.
  Interventions: Other: Peanut Consumption

INTERVENTIONS:
Other: High Intensity Interval Training — Subjects will exercise according the the high intensity aerobic interval training regiment four times a week for four weeks
  Other Names: Aerobic Exercise
  Arms: High Intensity Interval Training then Peanut Consumption
Other: Peanut Consumption — Subjects will consume peanuts twice a day to replace 20% of their daily caloric intake for four weeks.
  Arms: Peanut Consumption then High Intensity Interval Training

SUMMARY:
This study will enroll and randomly assign 30 sedentary, healthy overweight men and women to two groups. Participants will either start by consuming peanuts for 4 weeks, and then go on to exercise at high intensity intervals (HIIT) for 4 weeks, or the reverse order. The study will test and compare the effect of peanuts and exercise on inflammation and heart rate variability as indicators of heart health. Specifically, the study will measure inflammation in the blood because there is evidence that higher inflammation is found in heart disease patients. There is also evidence that inflammation is related to death as a result of heart disease in healthy individuals. Finally, there are ongoing trials targeting these markers to improve heart health. The study hypothesizes that peanuts and exercise will reduce inflammation. It is also expected to find less inflammation because exercise and peanut consumption activate a part of the nervous system that has been shown to cause a similar effect.

Additionally, previous studies show that inflammation involves the mitochondria in the cell, the part of the cell that produces energy. For this reason, it is expected that exercise and peanuts will cause changes in the mitochondria. The study will test and compare mitochondrial activity in response to peanut consumption and exercise.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Of either sex,
  2. age 21-45 years
  3. English-speaker
  4. Overweight or obese
  5. sedentary
* EXCLUSION CRITERIA

  1. Cardiovascular disease
  2. Uncontrolled high blood pressure (blood pressure ≥ 140/90). Individuals with controlled hypertension (i.e. under medical treatment) and blood pressure lower than 140/90 will not be excluded.
  3. Current or recent (evidence of disease x 5 years) non-skin neoplastic disease or melanoma. Prostatic carcinoma will not be grounds for exclusion.
  4. Active hepatic disease (not a history of hepatitis) or primary renal disease requiring dialysis, primary untreated endocrine diseases, e.g., Cushing's disease or primary hypothalamic failure or insulin dependent diabetes (Type I or II).
  5. HIV infection
  6. Pregnant or lactating (participation allowed 3 months after ceasing lactation).
  7. Medications that alter inflammation or autonomic nervous system activity.
  8. Any history of psychosis or ECT
  9. Psychotic disorder (lifetime)
  10. Current or recent (past 5 years) Major Depressive Disorder, Bipolar Disorder, or Anxiety disorder
  11. Current or recent (within past 12 months) alcohol or substance abuse or dependence. Recent use (past month) of recreational drugs.
  12. Probiotic and dietary supplements that affect inflammation or the ANS
  13. Physically active
  14. Peanut allergy in subject or in family of subject. Subjects who are unsure of their allergy status will be excluded.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard p Sloan, PhD, Principal Investigator — CUMC/NYSPI
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
data will be made available in June 2018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study terminated at early stage due to poor enrollment
Groups:
- High Intensity Interval Training First Then Peanut Consumption: Participants will engage in high intensity interval training first then peanut consumption
  High intensity interval training:
  4 training sessions per week over a 4-week period, with 24hour rest-periods between each training day. Each session begins with a 3 min low intensity warm-up, and then participants exercise as rapidly as they can for 20 seconds, aiming to reach 85% of their maximum heart rate as established during the submaximal cardiopulmonary exercise testing. This 20 second period is followed by 40 seconds of low intensity exercise.
- Peanut Consumption First Then High Intensity Interval Training: Peanut consumption first then high intensity interval Training
  Peanut Consumption:
  Subjects will consume peanuts twice a day to replace 20% of their daily caloric intake for four weeks.
  Daily caloric intake will be estimated using data from 24hr recalls, the Miflin-St. Jeor equation, and stress/activity factors. Peanuts replaces protein and fat containing foods so that the daily caloric intake will not differ from diet. To assess compliance, participants will be asked to bring back the empty, numbered peanut packets by the end of every week and will be given new packets weekly. Subjects will be informed that they will be randomly assessed weekly for compliance; they will be asked to provide details of when and where they consumed their packets the previous day.
Period: First Sequence (4 Weeks)
Arm/Group | High Intensity Interval Training First Then Peanut Consumption | Peanut Consumption First Then High Intensity Interval Training
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Washout (4 Weeks)
Arm/Group | High Intensity Interval Training First Then Peanut Consumption | Peanut Consumption First Then High Intensity Interval Training
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Second Sequence (4 Weeks)
Arm/Group | High Intensity Interval Training First Then Peanut Consumption | Peanut Consumption First Then High Intensity Interval Training
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- High Intensity Interval Training First Then Peanut Consumption: High intensity interval training first then peanut consumption
  High intensity interval training:
  4 training sessions per week over a 4-week period, with 24hour rest-periods between each training day. Each session begins with a 3 min low intensity warm-up, and then participants exercise as rapidly as they can for 20 seconds, aiming to reach 85% of their maximum heart rate as established during the submaximal cardiopulmonary exercise testing. This 20 second period is followed by 40 seconds of low intensity exercise.
- Total: Total of all reporting groups
Arm/Group | High Intensity Interval Training First Then Peanut Consumption | Peanut Consumption First Then High Intensity Interval Training | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (0) | 25 (0) | 31.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Plasma Levels of Pro-inflammatory Cytokines (IL-6 and TNF-α)
Description: cytokines (IL-6 and TNF-α) will be collected from blood samples
Time Frame: at study entry
Population: Study was terminated due to poor enrollment. No data was analyzed.
Groups:
- High Intensity Interval Training - Aerobic Exercise: Participants will engage in 4 training sessions per week over a 4-week period, with 24 hour rest-periods between each training day. Each session begins with a 3 min low intensity warm-up, and then participants exercise as rapidly as they can for 20 seconds, aiming to reach 85% of their maximum heart rate as established during the submaximal cardiopulmonary exercise testing. This 20 second period is followed by 40 seconds of low intensity exercise.
  High Intensity Interval Training: Subjects will exercise according the the high intensity aerobic interval training regiment four times a week for four weeks
- Peanut Consumption: Regular daily caloric intake of each subject will be estimated using data from 24hr recalls, the Miflin-St. Jeor equation, and stress/activity factors. Participants will consume dry roasted, unsalted peanuts equivalent to approximately 10% of daily energy intake twice (total=20% total), which will range from 400kcal to 600 kcal, which corresponds to about 2.4 oz to 3.6 oz. Peanuts will replace protein and fat containing foods so that the daily caloric intake will not differ from participants' typical diet. To assess compliance, participants will be asked to bring back the empty, numbered peanut packets by the end of every week and will be given new packets weekly.Subjects will be informed that they will be randomly assessed weekly for compliance; they will be asked to provide details of when and where they consumed their packets the previous day.
  Peanut Consumption: Subjects will consume peanuts twice a day to replace 20% of their daily caloric intake for four weeks.
Arm/Group | High Intensity Interval Training - Aerobic Exercise | Peanut Consumption
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | High Intensity Interval Training First Then Peanut Consumption | Peanut Consumption First Then High Intensity Interval Training
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03212144/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03212144/SAP_001.pdf
  • Informed Consent Form (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT03212144/ICF_002.pdf